CLINICAL TRIAL: NCT04348305
Title: Low-dose Hydrocortisone in Patients With COVID-19 and Severe Hypoxia - the COVID STEROID Trial
Brief Title: Hydrocortisone for COVID-19 and Severe Hypoxia
Acronym: COVID STEROID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Scandinavian Critical Care Trials Group (Other)
Collaborators: Rigshospitalet, Denmark (Other); Copenhagen Trial Unit, Center for Clinical Intervention Research (Other); University of Copenhagen (Other); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RH-ITA-008; 2020-001395-15 (EudraCT Number)
Record Dates: First submitted 2020-04-11; First posted 2020-04-16 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Covid-19; Hypoxia
MeSH Terms: conditions — COVID-19; Hypoxia | interventions — Hydrocortisone; hydrocortisone hemisuccinate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrocortisone (Experimental): Continuous intravenous infusion of hydrocortisone 200 mg over 24 hours (total 104 ml). The trial intervention will be given in addition to standard care.
  If continuous intravenous infusion is not possible, we will allow the use of bolus injection of the trial medication (50 mg (10 ml) every 6 hours).
  Interventions: Drug: Hydrocortisone
- Isotonic Saline (Placebo Comparator): Continuous intravenous infusion of matching isotonic saline (0.9%) placebo at a dose volume of 104 ml over 24 hours in addition to standard care (no corticosteroid treatment).
  If continuous intravenous infusion is not possible, we will allow the use of bolus injection of matching saline placebo (10 ml every 6 hours).
  Interventions: Drug: Sodium Chloride 9mg/mL

INTERVENTIONS:
Drug: Hydrocortisone — Continuous infusion: 200 mg (104 ml) every 24 hours, Bolus injections: 50 mg (10 ml) every 6 hours, Total treatment duration: 7 days
  Other Names: Solu-cortef
  Arms: Hydrocortisone
Drug: Sodium Chloride 9mg/mL — Continuous infusion: 104 ml every 24 hours, Bolus injections: 10 ml every 6 hours, Total treatment duration: 7 days
  Other Names: Isotonic saline
  Arms: Isotonic Saline

SUMMARY:
We aim to assess the benefits and harms of low-dose hydrocortisone in patients with COVID-19 and severe hypoxia.

DETAILED DESCRIPTION:
Background: Severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) has caused a pandemic of coronavirus disease (COVID-19) with many patients developing severe hypoxic respiratory failure. Many patients have died, and healthcare systems in several countries have been or will be overwhelmed because of a surge of patients needing hospitalisation and intensive care. There is no proven treatment for COVID-19; the care is supportive, including respiratory and circulatory support. For other patient groups with similar critical illness (acute respiratory disease syndrome and septic shock), corticosteroids are used because they reduce the duration of mechanical ventilation, length of stay in the intensive care unit, and potentially also mortality. Corticosteroids have been used in some patients with COVID-19, but the recommendations in clinical guidelines differ; some suggest their use, others against.

Objectives: We aim to assess the effects of low-dose intravenous hydrocortisone on the number of days alive without life-support in adult patients with COVID-19 and severe hypoxia.

Design: Multicentre, parallel-group, centrally randomised, stratified, blinded, clinical trial.

Population: Adult patients with documented COVID-19 receiving at least 10 L/min of oxygen independent of delivery system OR mechanical ventilation.

Experimental intervention: Continuous IV infusion of hydrocortisone 200 mg daily will be given for 7 days in addition to standard care.

Control intervention: Continuous IV infusion of matching placebo (0.9% saline) will be given in addition to standard care (no corticosteroids).

Outcomes: The primary outcome is days alive without life support (i.e. mechanical ventilation, circulatory support, or renal replacement therapy) at day 28. Secondary outcomes are serious adverse reactions (i.e. anaphylactic reaction to hydrocortisone, new episode of septic shock, invasive fungal infection or clinically important gastrointestinal bleeding); days alive without life support at day 90; days alive and out of hospital at day 90; all-cause mortality at day 28, day 90 and 1 year; and health-related quality of life at 1 year.

Sample size: A total of 1000 participants will be randomised in order to detect a 15% relative reduction in 28-day mortality combined with a 10% reduction in time on life support among the survivors with a power of 85%.

ELIGIBILITY:
Inclusion Criteria:

All the following criteria must be fulfilled:

* Aged 18 years or above AND
* Confirmed SARS-CoV-2 (COVID-19) requiring hospitalisation AND
* Use of one of the following:

  * Invasive mechanical ventilation OR
  * Non-invasive ventilation or continuous use of continuous positive airway pressure (CPAP) for hypoxia OR
  * Oxygen supplementation with an oxygen flow of at least 10 L/min independent of delivery system

Exclusion Criteria:

We will exclude patients who fulfil any of the following criteria:

* Use of systemic corticosteroids for any other indication than COVID-19
* Invasive mechanical ventilation for more than 48 hours
* Invasive fungal infection
* Fertile woman (< 60 years of age) with positive urine human gonadotropin (hCG) or plasma-hCG
* Known hypersensitivity to hydrocortisone
* A patient for whom the clinical team has decided not to use invasive mechanical ventilation
* Previously randomised into the COVID STEROID trial
* Informed consent not obtainable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-04-17 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2021-09-08 (Actual)

PRIMARY OUTCOMES:
Days alive without life support at day 28 | Day 28 after randomisation
  Days alive without life support (i.e. invasive mechanical ventilation, circulatory support or renal replacement therapy) from randomisation to day 28

SECONDARY OUTCOMES:
All-cause mortality at day 28 | Day 28 after randomisation
  Death from all causes
Days alive without life support at day 90 | Day 90 after randomisation
  Days alive without life support (i.e. invasive mechanical ventilation, circulatory support or renal replacement therapy) from randomisation to day 90
All-cause mortality at day 90 | Day 90 after randomisation
  Death from all causes
Number of participants with one or more serious adverse reactions | Day 14 after randomisation
  Defined as new episodes of septic shock, invasive fungal infection, clinically important GI bleeding or anaphylactic reaction
Days alive and out of hospital at day 90 | Day 90 after randomisation
  Number of days alive and out of hospital not limited to the index admission
All-cause mortality at 1 year after randomisation | 1 year after randomisation
  Death from all causes
Health-related quality of life at 1 year | 1 year after randomisation
  Assessed by EQ-5D-5L
Health-related quality of life at 1 year | 1 year after randomisation
  Assessed by EQ-VAS

CONTACTS AND LOCATIONS:
Overall Officials: Anders Perner, MD, PhD, Study Chair — Rigshospitalet, Denmark
Locations (14):
- Denmark (14):
  - Aarhus University Hospital - Dept of Intensive care, Aarhus
  - Rigshospitalet, Copenhagen
  - Dept of Infectious diseases, Rigshospitalet, Copenhagen
  - Herlev Hospital - Dept. of Intensive Care, Herlev
  - North Zealand Hospital, Hillerød
  - Hvidovre Hospital - Dept of Infectious diseases, Hvidovre
  - Hvidovre Hospital - Dept of Intensive Care, Hvidovre
  - Hvidovre Hospital - Dept of Pulmonary Medicine, Hvidovre
  - Kolding Hospital, Kolding
  - Køge Hospital, Køge
  - Dept of Intensive Care, Odense University Hospital, Odense
  - Roskilde Hospital, Roskilde
  - Slagelse Hospital, Slagelse
  - Viborg Hospital, Viborg

IPD SHARING:
Plan to Share IPD: Yes
Fully de-identified IPD will be shared after the approval by the the trial management committee
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediate sharing of protocol, SAP and ICF. CSR will be shared no later than 6 months after last-patient-last-visit
Access Criteria: Contact to the trial management committee
URL: http://www.cric.nu/covid-steroid-trial/

REFERENCES:
- [Derived] Munch MW, Granholm A, Kjaer MN, Aksnes TS, Solling CG, Christensen S, Perner A. Long-term mortality and health-related quality of life in the COVID STEROID trial. Acta Anaesthesiol Scand. 2022 Apr;66(4):543-545. doi: 10.1111/aas.14029. Epub 2022 Feb 3. No abstract available. PMID 35067914
- [Derived] Munch MW, Meyhoff TS, Helleberg M, Kjaer MN, Granholm A, Hjortso CJS, Jensen TS, Moller MH, Hjortrup PB, Wetterslev M, Vesterlund GK, Russell L, Jorgensen VL, Kristiansen KT, Benfield T, Ulrik CS, Andreasen AS, Bestle MH, Poulsen LM, Hildebrandt T, Knudsen LS, Moller A, Solling CG, Brochner AC, Rasmussen BS, Nielsen H, Christensen S, Strom T, Cronhjort M, Wahlin RR, Jakob SM, Cioccari L, Venkatesh B, Hammond N, Jha V, Myatra SN, Jensen MQ, Leistner JW, Mikkelsen VS, Svenningsen JS, Laursen SB, Hatley EV, Kristensen CM, Al-Alak A, Clapp E, Jonassen TB, Bjerregaard CL, Osterby NCH, Jespersen MM, Abou-Kassem D, Lassen ML, Zaabalawi R, Daoud MM, Abdi S, Meier N, la Cour K, Derby CB, Damlund BR, Laigaard J, Andersen LL, Mikkelsen J, Jensen JLS, Rasmussen AH, Arnerlov E, Lykke M, Holst-Hansen MZB, Tostesen BW, Schwab J, Madsen EK, Gluud C, Lange T, Perner A. Low-dose hydrocortisone in patients with COVID-19 and severe hypoxia: The COVID STEROID randomised, placebo-controlled trial. Acta Anaesthesiol Scand. 2021 Nov;65(10):1421-1430. doi: 10.1111/aas.13941. Epub 2021 Sep 20. PMID 34138478
- See also: Related Info — http://www.cric.nu/covid-steroid-trial/